CLINICAL TRIAL: NCT02584166
Title: Intervention of Psychological and Ethical Professionals of Human Science in Obstetrical Morbidity and Mortality Conferences
Brief Title: Intervention of Psychological and Ethical Professionals of Human Science in Obstetrical Morbidity and Mortality Conferences (OPERA)
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50791
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Newborns
Keywords: Morbidity; Mortality; conferences; human science

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention group: 38 maternity units with allocated to the intervention group: coordinating team disseminated protocols related to the management of cases, and organized mortality morbidity conferences (MMC) in each unit with staff concerned. These MMC were realized by the same outside medical binomial composed of a midwife and an obstetrician (outreach visit with a leader ship). Among the 38 maternity units, MMC were performed with the medical binomial and professionals of human science in 20 units to identify the defense mechanisms manifested by medical staff which could disturb the decision making. In the others 18 units, MMC were performed with only the outside medical binomial. Coordinating team defined with teams the area of improvement before each MMC. 3 or 4 MMC were performed according to their activity.
  Interventions: Behavioral: multifaceted program
- Control group: No intervention in 57 maternity units

INTERVENTIONS:
Behavioral: multifaceted program — This program present two steps : a first step to revise protocols related to the management of cases (between M5 and M8) and a second step after M8 et M 26, with morbimortality conferences organized every trimester to analyze management with the staff.
  Groups: Intervention group

SUMMARY:
This cluster-randomised controlled trial will test the hypothesis that a multifaceted program with psychological intervention in morbidity mortality conferences (MMC) improve care quality and reduce the rate of morbidity mortality perinatal in diverse obstetric care settings.

ELIGIBILITY:
Inclusion Criteria:

* all newborns born between 1er october 2008 and 30 November 2010 (minimum : 22 weeks of gestation)

Exclusion Criteria:

* newborns died in context of abortion

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns born between 1er october 2008 and 30 November 2010 (in one of the 95 maternity units which belongs to one of the 5 perinatal networks).
Sampling Method: Non-Probability Sample
Enrollment: 4929 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the rate of non conform management of morbidity and mortality cases | at 26th month
  Comparison in the two groups

SECONDARY OUTCOMES:
the rate of avoidable mortality and morbidity cases | at 26th month
  Comparison in the two groups
the incidence of mortality and morbidity among number of births | at 26th month
  Comparison in the two groups

REFERENCES:
- [Derived] Dupont C, Winer N, Rabilloud M, Touzet S, Branger B, Lansac J, Gaucher L, Duclos A, Huissoud C, Boutitie F, Rudigoz RC, Colin C; OPERA group. Multifaceted intervention to improve obstetric practices: The OPERA cluster-randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2017 Aug;215:206-212. doi: 10.1016/j.ejogrb.2017.06.026. Epub 2017 Jun 19. PMID 28649035